CLINICAL TRIAL: NCT00223587
Title: Study to Investigate the Effects of Seasonal Allergic Rhinitis on Over-the-Road Driving Performance and Memory Functioning
Brief Title: Seasonal Allergic Rhinitis and Driving Ability
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Joris C Verster, Utrecht University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04/089-E
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: driving; memory
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 1 week of treatment discontinuation
  Interventions: Other: 1 week of treatment discontinuation

INTERVENTIONS:
Other: 1 week of treatment discontinuation — 1 week of treatment discontinuation during allergic rhinitis season

SUMMARY:
On-the-road driving performance of untreated seasonal allergic rhinitis patients during the allergic season (exposed) is compared to driving performance outside the allergic season (in winter, not-exposed).

DETAILED DESCRIPTION:
This study was set-up to examine whether untreated seasonal allergic rhinitis has an effect on driving ability. In addition to the driving tests, patients perform a memory test in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with seasonal allergic rhinitis
* a valid driver's licence
* written informed consent
* a T5SS score >8 during the allergic season and <3 in winter

Exclusion Criteria:

* use of medication or medical conditions that are known to affect driving ability
* associated ENT disease or asthma

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Driving test: Standard Deviation of Lateral Position (SDLP, cm); i.e. the weaving of the car [after 1 week of treatment discontinuation] | allergic season and winter

SECONDARY OUTCOMES:
Other driving test parameters: standard deviation of speed, mean speed, meal lateral position [after 1 week of treatment discontinuation] | allergic season and winter
Memory test: immediate and delayed recall, delayed recognition [after 1 week of treatment discontinuation] | allergic season and winter

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Volkerts, PhD, Study Director — Utrecht Institute for Pharmaceutical Sciences; Joris Verster, PhD, Principal Investigator — Utrecht Institute for Pharmaceutical Sciences
Locations (1):
- Utrecht Institute for Pharmaceutical Sciences, Utrecht, Netherlands